CLINICAL TRIAL: NCT04153162
Title: Non-Invasive Radiation Ablation for Septal Reduction in Patients With Hypertrophic Obstructive CardioMyopathy: First in Man Pilot Study
Brief Title: Non-Invasive Radiation Ablation in Patients With Hypertrophic CardioMyopathy: NIRA-HOCM
Acronym: NIRA-HOCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Barts Cardiovascular CTU (Queen Mary University of London) (Unknown); Barts Clinical Trial Unit (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIRA-HOCM 1.1
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic body radiation therapy (Experimental): In patients with HCM and refractory symptoms from LVOTO, stereotactic body radiation therapy will be delivered locally to relieve symptoms
  Interventions: Device: Stereotactic body radiation therapy

INTERVENTIONS:
Device: Stereotactic body radiation therapy — Stereotactic body radiation therapy delivered to reduce LVOTO in patients with HCM

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is a common disease of the heart which causes thickening of the heart muscle.

HCM primarily affects the muscle of the main pumping chamber of the heart (the left ventricle) and particularly the septum (this is the muscular wall which separates the right and left side of the heart). In a subgroup of patients, the thickened heart muscle at the septum prevents blood from leaving the heart during contraction (this is called obstruction). This form of the disease is called hypertrophic obstructive cardiomyopathy (HOCM).

HOCM is a common cause of shortness of breath, chest pain and dizzy spells. These symptoms are treated with tablets and if symptoms are uncontrolled, patients are often offered invasive treatment to get rid of some of the thick heart muscle and reduce obstruction. This is achieved either by:

1. open heart surgery (myectomy) where a surgeon cuts out the thick muscle
2. injection of alcohol to the thick heart muscle via a tube in the wrist or groin (alcohol septal ablation). The alcohol thins the heart muscle at the point of obstruction, mimicking the effects of myectomy.

Unfortunately, some patients are not suitable for both these procedures.

This study will test whether radiotherapy, usually used for the treatment of tumours, can be used to destroy the thick heart muscle at the point of obstruction safely and effectively. Study patients will be monitored following the procedure and the investigators plan to measure the levels of heart muscle thinning, reduction of obstruction and improvement in symptoms and importantly document any side effects.

Radiotherapy works by precisely targeting high energy X-rays (ionising radiation) at a specific area of the body with the aim of destroying abnormal tissue. CyberKnife is one of the latest radiotherapy delivery systems, which will deliver highly focussed and accurate radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Limiting, drug refractory symptoms secondary to left ventricular outflow tract obstruction
2. Previously failed invasive septal reduction therapy (ethanol septal ablation/surgical myectomy) or inability to perform invasive septal reduction due to increased risk/co-morbidities/anatomical considerations following specialist MDT review
3. A device (permanent pacemaker or implantable cardioverter defibrillator) in situ.
4. Ventricular septal thickness at site ablation ≥ 16mm.
5. Patient able to tolerate lying flat for one hour
6. High target-surrogacy of ICD/pacing lead for cardiac motion (from cardiac-gated MRI or cardiac-gated CT with the patient in pacing mode used for treatment)
7. Successful completion of ICD lead tip tracking test ("patient dummy run") with the patient in pacing mode used for treatment
8. Adult Patients aged 18 and over willing and able to give written informed consent

Exclusion Criteria:

1. New York Heart Association I-II
2. Canadian Cardiovascular Society class 1-2
3. Follow-up impossible (e.g. no fixed abode)
4. Weight of patient that exceeds the maximum limit of CMR table (170kg)
5. Subjects of childbearing potential unless βHCG negative and on contraception
6. Lack of cardiac device with anti-bradycardia pacing capabilities
7. Previous chest radiotherapy
8. Inability to provide informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Demonstrate acute (≤ 90 days) safety of non-invasive SBRT. | 90 days
  The primary safety endpoint is defined as serious adverse events (SAEs) that are possibly/probably/definitely related to study treatment, based on previously published data for expected invasive alcohol septal-ablation procedures.

SECONDARY OUTCOMES:
Assessment of MACE endpoints | 3, 6 and 12 months
  MACE = death, heart failure, myocardial infarction and stroke
Change in aortic valve and mitral valve function | 3, 6 and 12 months
  Echocardiography assessed aortic and mitral valve function
Left anterior descending artery patency | 12 months
  Patency of left anterior descending artery with cardiac CT
Presence of radiation pneumonitis | 12 months
  Presence of radiation pneumonitis on CT
Development of complete heart block, atrial or ventricular arrhythmias | 3, 6 and 12 months
  Cardiac device (ICD or pacemaker) check
Change in LVOT gradient | 3, 6 and 12 months
  Assessed with transthoracic echocardiography using same loading conditions as baseline
Change in functional class | 6 and 12 months
  Change in NYHA and CCS class from baseline
Change in frequency of syncope and pre-syncope | 6 and 12 months
  Baseline to 6 and 12 months
Change in exercise capacity | 6 and 12 months compared to Baseline
  6 minute Walk Test
Change in health status | 6 and 12 months compared to Baseline
  EQ-5D-5L
Troponin T elevation | 1,2,3 days post ablation
  Measurement of Trop T
Change in LV wall thickness | 6 months
  CMR assessed thickness
Left ventricular ejection fraction (LVEF) | 3, 6 and 12 months
  Measured on echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Costas O'Mahony, FRCP, MD, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Heart Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No